CLINICAL TRIAL: NCT06606821
Title: The Effects of Tirzepatide on Coronary Plaque Lipid Content and Myocardial Microvascular Function in Overweight and Obese People With Coronary Disease - The IDEAL-COR Study
Brief Title: The Effects of Tirzepatide in People With Overweight/Obesity and Coronary Artery Disease
Acronym: IDEAL-COR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tina Vilsbøll (Other)
Responsible Party: Sponsor-Investigator, Tina Vilsbøll, Professor, MD DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-505270-15-00; 2023-505270-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-04; First posted 2024-09-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; Coronary Microvascular Dysfunction; Overweight or Obesity; Stable Angina Pectoris; Chronic Coronary Artery Disease; Atherosclerosis Cardiovascular Disease
Keywords: NIRS; IVUS; GLP-1; Tirzepatide; Intravascular imagining; Stable Angina Pectoris
MeSH Terms: conditions — Coronary Artery Disease; Overweight; Obesity; Angina, Stable | interventions — Tirzepatide; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide (Experimental): Tirzepatide is administered sc. once-weekly.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Placebo is administered sc. once-weekly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Investigational drug will be administered as a sc. injection once-weekly.
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Placebo containing the same excipients and volume as the active treatment arm but without tirzepatide will be administered as a sc. injection once-weekly.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate, as a proof-of-principle, long-term (52 weeks) effects of tirzepatide once-weekly vs. placebo on changes in coronary plaque composition and progression (assessed by NIRS), plaque burden (assessed by IVUS) and microvascular function (assessed by invasively measured CFR) in overweight and obese individuals with stable coronary artery disease (CAD). In addition, the objective of a baseline cross-sectional sub-study is to explore potential metabolic and cardiovascular (CV) predictors for high arteriosclerotic plaque burden in overweight and obese individuals and to establish a cohort for future research projects.

DETAILED DESCRIPTION:
The anti-atherogenic effect of tirzepatide has been studied in preclinical studies and seems to involve mechanisms related to a reduction in vascular inflammation and lipid accumulation. Any direct anti-atherogenic effect of tirzepatide may potentially reduce the incidence of major cardiovascular endpoints in individuals with overweight or obesity. As a proof of principle, it would be of scientific and clinical interest to explore the anti-atherogenic effect of tirzepatide in humans. IVUS-NIRS imaging is uniquely suited for this purpose, as it makes it possible to detect changes in not only atheroma burden by IVUS but also to detect progression within the plaques in the lipidic/necrotic core component by NIRS. LCBItotal allows for consecutive detection of small changes in the same individual, which is pivotal to explore the supposed antiatherogenic mechanism of tirzepatide with enough statistical power.

The investigators hypothesize that once-weekly sc. tirzepatide can reduce coronary lipid accumulation in the arterial wall and the progression of atheromatosis in individuals with overweight or obesity and established high-risk atherosclerosis. The investigators aim to investigate this hypothesis in a proof-of-principle study by investigating the change in coronary plaque composition in individuals with overweight or obesity and coronary artery disease (CAD) with high-risk characteristics by NIRS imaging randomised to 52-week treatment with tirzepatide or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent
* BMI equal to or above 27 kg/m2
* Age 18 years or older
* Referred to coronary angiogram (CAG) due to stable angina
* Coronary atheromatosis by angiography (obstructive or non-obstructive)
* LCBI4mm >200 by NIRS in a vessel not subjected to coronary intervention

Exclusion Criteria:

* History of diabetes or HbA1c ≥48 mmol/mol (6.5%) at baseline
* Treatment with Glucagon-Like Peptide-1 Receptor Agonists (GLP-1RA)
* History of coronary artery bypass surgery (CABG)
* Planned CV intervention (including percutaneous coronary intervention, cardiac surgery or transcatheter valve intervention) at time of randomisation
* History of heart failure New York Heart Association (NYHA) class III or IV
* Left ventricular ejection fraction (LVEF) ≤35%
* eGFR <30 ml/min/1.53 m2
* History of pancreatitis or plasma amylase >2 times upper normal limit
* Impaired hepatic function at baseline (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times the upper limit of normal)
* Pregnancy, planned pregnancy or breastfeeding
* Family or history of multiple endocrine neoplasia (MEN) type 2 or familial medullary thyroid carcinoma (FMTC)
* Hypersensitivity to the active substance (Tirzepatide) or to any of the excipients
* Left main stenosis (≥50% diameter or haemodynamically significant)
* Chronic total occlusion of any major coronary vessel
* Multi-vessel disease or complex anatomy potentially requiring coronary bypass surgery
* Coronary anatomy or pathology precluding the safe performance of intravascular imaging in all major coronary arteries not subjected to intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Lipid core burden index | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Lipid core burden index of the three major coronary vessels (LCBItotal) measured by NIRS imaging.

SECONDARY OUTCOMES:
Percent atheroma volume (PAV) | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Total coronary plaque burden measured by coronary IVUS imaging assessed by Percent atheroma volume (PAV)
Number of high-risk coronary lesion | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Number of high-risk coronary lesions characterized by maximum lipid core burden index of a 4 mm examined vessel (maxLCBI4mm) ≥325 and plaque burden ≥70%
Coronary flow reserve | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Coronary flow reserve (CFR) assessed by invasive coronary thermodilution technique during coronary angiogram measures the blood flow in the epicardial arteries and the microvasculature.

OTHER OUTCOMES:
Plasma lipid profile | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Total cholesterol (TC) Triglyceride (TG) High-density lipoprotein cholesterol (HDL-C) LDL-C
Markers of inflammation | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  High-sensitive C-reactive protein (hsCRP) Interleukin-6 (IL-6)
Left ventricular systolic and diastolic function assessed by echocardiography: | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Global longitudinal strain (GLS) measured by speckle tracking E/e' measured by tissue-Doppler
Body composition assessed by DXA scan: | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Regional visceral adipose tissue (VAT) Bone density
Urine markers of oxidative stress | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  8-oxo-7,8-dihydro2´-deoxyguanosine (8-oxodG) 8-oxo-7,8-dihydroguanosine (8-oxoGuo)
Myocardial work | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Assessed by pressure-strain loop analysis derived from speckle-tracking echocardiography
Seattle Angina Questionnaire-7 | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Seattle Angina Questionnaire-7 (SAQ-7) measures health status in patients with coronary artery disease. The SAQ-7 generates a summary score (scale 0-100, 100 = full health, 0 = worst health).
Thromboelastography | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Thromboelastography is a viscoelastic hemostatic assay that measures the global viscoelastic properties of whole blood clot formation under low shear stress
  The following parameters will be measured:
  * R value = reaction time (min)
  * K = kinetics (min)
  * alpha = angle (degrees)
  * MA = maximum amplitude (mm) Represents the ultimate strength of the fibrin clot; i.e. overall stability of the clot
  * LY30 = amplitude at 30 minutes (%) Percentage decrease in amplitude at 30 minutes post-MA
EuroQoL 5-Dimension 5-Level | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  The EuroQoL 5-Dimension 5-Level (EQ-5D-5L) is questionnaire of 5 health dimensions - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression - and includes 5 response categories of no problem, slight problems, moderate problems, severe problems, and extreme problems. The 5 responses give a health state or profile represented by a 5-digit number (for example, 12231) corresponding to response categories reported by patients for successive dimensions, beginning with mobility. Health states are scored to give the EQ-5D-5L index using a scoring algorithm from a value set derived from valuation tasks typically undertaken with general population samples. Index scores range from -0.59 to 1; 1 is the best possible health state.
Liver stiffness measurement | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Liver Stiffness Measurement (LSM): This measurement is performed using a technology called Fibroscan. It measures the stiffness or hardness of the liver, which correlates with the degree of liver fibrosis (scarring). The result is expressed in kilopascals (kPa). Normal liver stiffness values typically range from 2 to 7 kPa, with higher values indicating more severe fibrosis.
Controlled Attenuation Parameter | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Controlled Attenuation Parameter (CAP): This measurement is performed using a technology called Fibroscan. This measures the amount of fat in the liver, known as steatosis. The CAP score is expressed in decibels per meter (dB/m) and ranges from 100 to 400 dB/m. Higher CAP scores indicate greater levels of liver fat.
Homeostatic Model Assessment for Insulin Resistance | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Homeostatic model assessment of insulin resistance (HOMA-IR) evaluates systemic insulin resistance. HOMA-IR is calculated using fasting blood glucose and fasting insulin levels. The formula for HOMA-IR is: HOMA-IR = (Fasting Insulin uU/mL * Fasting Glucose mmol/L)/22.5
  HOMA-IR values between 0.5 and 1.4 are considered normal. ≥1.9 are indicative of early insulin resistance, and ≥2.9 indicate insulin resistance.
Fibrosis-4 score | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Fibrosis-4 (FIB-4) score is a non-invasive scoring system used to estimate the amount of liver fibrosis in individuals. The score is calculated using the following formula:
  FIB-4 = (Age * aspartate aminotransferase level U/L )/(Platelet count 10^9/L * squareroot(alanine aminotransferase level U/L ))
  The resulting score helps to stratify patients into different risk categories for liver fibrosis Low risk: FIB-4 under 1.3 Intermediate risk: FIB-4 between 1.3 and 2.67 High risk: FIB-4 above 2.67
Glycaemic profile | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Glycaemic variability measured by continuous glucose monitoring (CGM) Fasting plasma glucose (FPG) Glycated haemoglobin A1c (HbA1c)
Change in glycaemic variability | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Glycaemic variability measured by continuous glucose monitoring (CGM) refers to the fluctuations in blood glucose levels over time.
  The following metrics are used to quantify glycaemic variability:
  Standard Deviation (SD): Measures the dispersion of glucose values around the mean.
  Coefficient of Variation (CV): The ratio of the standard deviation to the mean glucose level, expressed as a percentage.
  Mean Amplitude of Glycemic Excursions (MAGE): Captures the average of the absolute differences between consecutive peaks and nadirs in glucose levels.
  Continuous Overlapping Net Glycemic Action (CONGA): Measures the variability of glucose levels over a specified period.
Change in fasting plasma glucose | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Fasting plasma glucose (FPG)
Change in glycated haemoglobin A1c | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo:
  Glycated haemoglobin A1c (HbA1c)
Index of microcirculatory resistance | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo
  Index of microcirculatory resistance (IMR) assessed by coronary thermodilution technique during coronary angiogram
Resistive Reserve Ratio | Between-group difference in change from baseline to week 52 in participants treated with tirzepatide vs placebo
  Resistive Reserve Ratio (RRR) assessed by coronary thermodilution technique during coronary angiogram is a measure used to evaluate the vasodilatory capacity of the coronary microvasculature.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD, DMSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (3):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Gentofte Municipality
  - Steno Diabetes Center Copenhagen, Herlev

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the clinical trial, after de-identification will be available in accordance with Danish data regulations.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 1 year after the end of the trial and publication of the primary outcomes, and will be available for 24 months.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal. Proposals should be directed to Prof. Tina Vilsbøll, MD DMSc, at tina.vilsboell.01@regionh.dk. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Jastreboff AM, Aronne LJ, Ahmad NN, Wharton S, Connery L, Alves B, Kiyosue A, Zhang S, Liu B, Bunck MC, Stefanski A; SURMOUNT-1 Investigators. Tirzepatide Once Weekly for the Treatment of Obesity. N Engl J Med. 2022 Jul 21;387(3):205-216. doi: 10.1056/NEJMoa2206038. Epub 2022 Jun 4. PMID 35658024
- [Background] Stoner MCD, Bhushan NL, Maragh-Bass AC, Mitchell JT, Riggins L, Walker M, LeMasters K, Reese B, Dearing A, Debnam S, Golin C, Lightfoot AF, Pettifor A. Using Participatory Methods to Assess PrEP Interest and Uptake Among Young People Living in the Southeastern US: A Mixed Methods Assessment. AIDS Behav. 2022 May;26(5):1672-1683. doi: 10.1007/s10461-021-03519-y. Epub 2021 Nov 1. PMID 34724592
- [Background] Coskun T, Sloop KW, Loghin C, Alsina-Fernandez J, Urva S, Bokvist KB, Cui X, Briere DA, Cabrera O, Roell WC, Kuchibhotla U, Moyers JS, Benson CT, Gimeno RE, D'Alessio DA, Haupt A. LY3298176, a novel dual GIP and GLP-1 receptor agonist for the treatment of type 2 diabetes mellitus: From discovery to clinical proof of concept. Mol Metab. 2018 Dec;18:3-14. doi: 10.1016/j.molmet.2018.09.009. Epub 2018 Oct 3. PMID 30473097
- [Background] Frias JP, Nauck MA, Van J, Kutner ME, Cui X, Benson C, Urva S, Gimeno RE, Milicevic Z, Robins D, Haupt A. Efficacy and safety of LY3298176, a novel dual GIP and GLP-1 receptor agonist, in patients with type 2 diabetes: a randomised, placebo-controlled and active comparator-controlled phase 2 trial. Lancet. 2018 Nov 17;392(10160):2180-2193. doi: 10.1016/S0140-6736(18)32260-8. Epub 2018 Oct 4. PMID 30293770
- [Background] Frias JP, Davies MJ, Rosenstock J, Perez Manghi FC, Fernandez Lando L, Bergman BK, Liu B, Cui X, Brown K; SURPASS-2 Investigators. Tirzepatide versus Semaglutide Once Weekly in Patients with Type 2 Diabetes. N Engl J Med. 2021 Aug 5;385(6):503-515. doi: 10.1056/NEJMoa2107519. Epub 2021 Jun 25. PMID 34170647
- [Background] Kristensen SL, Rorth R, Jhund PS, Docherty KF, Sattar N, Preiss D, Kober L, Petrie MC, McMurray JJV. Cardiovascular, mortality, and kidney outcomes with GLP-1 receptor agonists in patients with type 2 diabetes: a systematic review and meta-analysis of cardiovascular outcome trials. Lancet Diabetes Endocrinol. 2019 Oct;7(10):776-785. doi: 10.1016/S2213-8587(19)30249-9. Epub 2019 Aug 14. PMID 31422062
- [Background] Caruso I, Cignarelli A, Giorgino F. Heterogeneity and Similarities in GLP-1 Receptor Agonist Cardiovascular Outcomes Trials. Trends Endocrinol Metab. 2019 Sep;30(9):578-589. doi: 10.1016/j.tem.2019.07.004. Epub 2019 Aug 7. PMID 31401015
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 6. Glycemic Targets: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S97-S110. doi: 10.2337/dc23-S006. PMID 36507646
- [Background] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Background] Hernandez AF, Green JB, Janmohamed S, D'Agostino RB Sr, Granger CB, Jones NP, Leiter LA, Rosenberg AE, Sigmon KN, Somerville MC, Thorpe KM, McMurray JJV, Del Prato S; Harmony Outcomes committees and investigators. Albiglutide and cardiovascular outcomes in patients with type 2 diabetes and cardiovascular disease (Harmony Outcomes): a double-blind, randomised placebo-controlled trial. Lancet. 2018 Oct 27;392(10157):1519-1529. doi: 10.1016/S0140-6736(18)32261-X. Epub 2018 Oct 2. PMID 30291013
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Oh J, Teoh H, Leiter LA. Should C-reactive protein be a target of therapy? Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S155-60. doi: 10.2337/dc11-s211. No abstract available. PMID 21525448
- [Background] Howard G, Wagenknecht LE, Burke GL, Diez-Roux A, Evans GW, McGovern P, Nieto FJ, Tell GS. Cigarette smoking and progression of atherosclerosis: The Atherosclerosis Risk in Communities (ARIC) Study. JAMA. 1998 Jan 14;279(2):119-24. doi: 10.1001/jama.279.2.119. PMID 9440661
- [Background] Mundi S, Massaro M, Scoditti E, Carluccio MA, van Hinsbergh VWM, Iruela-Arispe ML, De Caterina R. Endothelial permeability, LDL deposition, and cardiovascular risk factors-a review. Cardiovasc Res. 2018 Jan 1;114(1):35-52. doi: 10.1093/cvr/cvx226. PMID 29228169
- [Background] Bai X, Yang X, Jia X, Rong Y, Chen L, Zeng T, Deng X, Li W, Wu G, Wang L, Li Y, Zhang J, Xiong Z, Xiong L, Wang Y, Zhu L, Zhao Y, Jin S. CAV1-CAVIN1-LC3B-mediated autophagy regulates high glucose-stimulated LDL transcytosis. Autophagy. 2020 Jun;16(6):1111-1129. doi: 10.1080/15548627.2019.1659613. Epub 2019 Sep 4. PMID 31448673
- [Background] Langheim S, Dreas L, Veschini L, Maisano F, Foglieni C, Ferrarello S, Sinagra G, Zingone B, Alfieri O, Ferrero E, Maseri A, Ruotolo G. Increased expression and secretion of resistin in epicardial adipose tissue of patients with acute coronary syndrome. Am J Physiol Heart Circ Physiol. 2010 Mar;298(3):H746-53. doi: 10.1152/ajpheart.00617.2009. Epub 2010 Jan 8. PMID 20061546
- [Background] Boren J, Chapman MJ, Krauss RM, Packard CJ, Bentzon JF, Binder CJ, Daemen MJ, Demer LL, Hegele RA, Nicholls SJ, Nordestgaard BG, Watts GF, Bruckert E, Fazio S, Ference BA, Graham I, Horton JD, Landmesser U, Laufs U, Masana L, Pasterkamp G, Raal FJ, Ray KK, Schunkert H, Taskinen MR, van de Sluis B, Wiklund O, Tokgozoglu L, Catapano AL, Ginsberg HN. Low-density lipoproteins cause atherosclerotic cardiovascular disease: pathophysiological, genetic, and therapeutic insights: a consensus statement from the European Atherosclerosis Society Consensus Panel. Eur Heart J. 2020 Jun 21;41(24):2313-2330. doi: 10.1093/eurheartj/ehz962. No abstract available. PMID 32052833
- [Background] Piche ME, Tchernof A, Despres JP. Obesity Phenotypes, Diabetes, and Cardiovascular Diseases. Circ Res. 2020 May 22;126(11):1477-1500. doi: 10.1161/CIRCRESAHA.120.316101. Epub 2020 May 21. PMID 32437302
- [Background] Kim SH, Despres JP, Koh KK. Obesity and cardiovascular disease: friend or foe? Eur Heart J. 2016 Dec 21;37(48):3560-3568. doi: 10.1093/eurheartj/ehv509. Epub 2015 Dec 18. PMID 26685971
- [Background] Hou J, Renigunta A, Konrad M, Gomes AS, Schneeberger EE, Paul DL, Waldegger S, Goodenough DA. Claudin-16 and claudin-19 interact and form a cation-selective tight junction complex. J Clin Invest. 2008 Feb;118(2):619-28. doi: 10.1172/JCI33970. PMID 18188451
- [Background] Nakamura K, Fuster JJ, Walsh K. Adipokines: a link between obesity and cardiovascular disease. J Cardiol. 2014 Apr;63(4):250-9. doi: 10.1016/j.jjcc.2013.11.006. Epub 2013 Dec 16. PMID 24355497
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Kang SJ, Mintz GS, Pu J, Sum ST, Madden SP, Burke AP, Xu K, Goldstein JA, Stone GW, Muller JE, Virmani R, Maehara A. Combined IVUS and NIRS detection of fibroatheromas: histopathological validation in human coronary arteries. JACC Cardiovasc Imaging. 2015 Feb;8(2):184-94. doi: 10.1016/j.jcmg.2014.09.021. Epub 2015 Jan 7. PMID 25577445
- [Background] Negi SI, Didier R, Ota H, Magalhaes MA, Popma CJ, Kollmer MR, Spad MA, Torguson R, Suddath W, Satler LF, Pichard A, Waksman R. Role of near-infrared spectroscopy in intravascular coronary imaging. Cardiovasc Revasc Med. 2015 Jul-Aug;16(5):299-305. doi: 10.1016/j.carrev.2015.06.001. Epub 2015 Jun 10. PMID 26242984
- [Background] Chen S, Okahara F, Osaki N, Shimotoyodome A. Increased GIP signaling induces adipose inflammation via a HIF-1alpha-dependent pathway and impairs insulin sensitivity in mice. Am J Physiol Endocrinol Metab. 2015 Mar 1;308(5):E414-25. doi: 10.1152/ajpendo.00418.2014. Epub 2014 Dec 23. PMID 25537494
- [Background] Otake H, Tanimura K, Sugizaki Y, Toba T, Kawamori H, Shinke T, Hirata KI. Effect of Alirocumab and Rosuvastatin or Rosuvastatin Alone on Lipid Core Plaque in Coronary Artery Disease Seen on Near-Infrared Spectroscopy Intravascular Ultrasound (ANTARES). Circ Rep. 2019 Jan 31;1(2):107-111. doi: 10.1253/circrep.CJ-18-0021. PMID 33693121
- [Background] Honda S, Sidharta SL, Shishikura D, Takata K, Di Giovanni GA, Nguyen T, Janssan A, Kim SW, Andrews J, Psaltis PJ, Worthley MI, Nicholls SJ. High-density lipoprotein cholesterol associated with change in coronary plaque lipid burden assessed by near infrared spectroscopy. Atherosclerosis. 2017 Oct;265:110-116. doi: 10.1016/j.atherosclerosis.2017.08.016. Epub 2017 Aug 31. PMID 28881268
- [Background] Kini AS, Vengrenyuk Y, Shameer K, Maehara A, Purushothaman M, Yoshimura T, Matsumura M, Aquino M, Haider N, Johnson KW, Readhead B, Kidd BA, Feig JE, Krishnan P, Sweeny J, Milind M, Moreno P, Mehran R, Kovacic JC, Baber U, Dudley JT, Narula J, Sharma S. Intracoronary Imaging, Cholesterol Efflux, and Transcriptomes After Intensive Statin Treatment: The YELLOW II Study. J Am Coll Cardiol. 2017 Feb 14;69(6):628-640. doi: 10.1016/j.jacc.2016.10.029. Epub 2016 Oct 29. PMID 27989886
- [Background] Kini AS, Baber U, Kovacic JC, Limaye A, Ali ZA, Sweeny J, Maehara A, Mehran R, Dangas G, Mintz GS, Fuster V, Narula J, Sharma SK, Moreno PR. Changes in plaque lipid content after short-term intensive versus standard statin therapy: the YELLOW trial (reduction in yellow plaque by aggressive lipid-lowering therapy). J Am Coll Cardiol. 2013 Jul 2;62(1):21-9. doi: 10.1016/j.jacc.2013.03.058. Epub 2013 May 1. PMID 23644090
- [Background] Biccire FG, Budassi S, Ozaki Y, Boi A, Romagnoli E, Di Pietro R, Bourantas CV, Marco V, Paoletti G, Debelak C, Sammartini E, Versaci F, Fabbiocchi F, Burzotta F, Pastori D, Crea F, Arbustini E, Alfonso F, Prati F. Optical coherence tomography-derived lipid core burden index and clinical outcomes: results from the CLIMA registry. Eur Heart J Cardiovasc Imaging. 2023 Mar 21;24(4):437-445. doi: 10.1093/ehjci/jeac110. PMID 35718858
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Trends in adult body-mass index in 200 countries from 1975 to 2014: a pooled analysis of 1698 population-based measurement studies with 19.2 million participants. Lancet. 2016 Apr 2;387(10026):1377-1396. doi: 10.1016/S0140-6736(16)30054-X. PMID 27115820
- [Background] Adair T, Lopez AD. The role of overweight and obesity in adverse cardiovascular disease mortality trends: an analysis of multiple cause of death data from Australia and the USA. BMC Med. 2020 Aug 4;18(1):199. doi: 10.1186/s12916-020-01666-y. PMID 32746822
- [Background] Patel D, Hamamdzic D, Llano R, Patel D, Cheng L, Fenning RS, Bannan K, Wilensky RL. Subsequent development of fibroatheromas with inflamed fibrous caps can be predicted by intracoronary near infrared spectroscopy. Arterioscler Thromb Vasc Biol. 2013 Feb;33(2):347-53. doi: 10.1161/ATVBAHA.112.300710. Epub 2013 Jan 3. PMID 23288155
- [Background] Virmani R, Kolodgie FD, Burke AP, Farb A, Schwartz SM. Lessons from sudden coronary death: a comprehensive morphological classification scheme for atherosclerotic lesions. Arterioscler Thromb Vasc Biol. 2000 May;20(5):1262-75. doi: 10.1161/01.atv.20.5.1262. No abstract available. PMID 10807742
- [Background] Lopez AD, Adair T. Is the long-term decline in cardiovascular-disease mortality in high-income countries over? Evidence from national vital statistics. Int J Epidemiol. 2019 Dec 1;48(6):1815-1823. doi: 10.1093/ije/dyz143. PMID 31378814
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Background] Raber L, Taniwaki M, Zaugg S, Kelbaek H, Roffi M, Holmvang L, Noble S, Pedrazzini G, Moschovitis A, Luscher TF, Matter CM, Serruys PW, Juni P, Garcia-Garcia HM, Windecker S; IBIS 4 (Integrated Biomarkers and Imaging Study-4) Trial Investigators (NCT00962416). Effect of high-intensity statin therapy on atherosclerosis in non-infarct-related coronary arteries (IBIS-4): a serial intravascular ultrasonography study. Eur Heart J. 2015 Feb 21;36(8):490-500. doi: 10.1093/eurheartj/ehu373. Epub 2014 Sep 2. PMID 25182248
- [Background] Weisbrod RM, Shiang T, Al Sayah L, Fry JL, Bajpai S, Reinhart-King CA, Lob HE, Santhanam L, Mitchell G, Cohen RA, Seta F. Arterial stiffening precedes systolic hypertension in diet-induced obesity. Hypertension. 2013 Dec;62(6):1105-10. doi: 10.1161/HYPERTENSIONAHA.113.01744. Epub 2013 Sep 23. PMID 24060894